CLINICAL TRIAL: NCT06881966
Title: The Effect of Omega-3 Fatty Acids in Patients With Rheumatoid Arthritis: A Study Protocol of a Double-blinded Randomized Controlled Trial
Brief Title: The Effect of Omega-3 Fatty Acids in Patients With Rheumatoid Arthritis
Acronym: omega3-RA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Charles Nicolle (Other)
Responsible Party: Principal Investigator, Selma Bouden, Assistant Doctor, Hopital Charles Nicolle
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ECR-OMG-2025-01; ECR-OMG-2025-01 (Other: Charles Nicolle Hospital)
Record Dates: First submitted 2025-03-07; First posted 2025-03-18 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: rheumatoid arthritis; omega3; supplementation; efficacy
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: All included patients will be randomized into two groups: an intervention group who will receive omega-3 supplementation and a control group who will receive placebo supplementation, over a period of 3 months.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- omega3 group (Experimental): Patients in the intervention group will consume 2 omega-3 capsules daily, which contain 36% and 24% of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), respectively, during a period of 3 months.
  The dose of omega-3 will be constant throughout the study period.
  Interventions: Dietary Supplement: Omega-3 Supplementation
- control group (Placebo Comparator): The control group will receive placebo supplementation, over a period of 3 months. The placebo capsules will be olive oil-based and will have the same visual as the omega-3 capsules. They will be developed by Vital Company. The dose of placebo will be constant throughout the study period.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 Supplementation — Patients in the intervention group will consume 2 omega-3 capsules (Omevie) daily, which contain 36% and 24% of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), respectively, during a period of 3 months.
  Arms: omega3 group
Other: Placebo — The control group who will receive placebo supplementation, over a period of 3 months.The placebo capsules will be olive oil-based and will have the same visual as the omega-3 capsules. They will be developed by Vital Company.
  Arms: control group

SUMMARY:
The aim of this double-blinded randomized controlled trial (RCT) was to assess the effect of omega-3 intake versus placebo among patients with RA on the primary outcome of disease activity, and the secondary outcomes of function, fatigue and sleep.

This is a prospective, comparative, randomized study, that will be conducted in a single centre (the Rheumatology Department of Charles Nicolle Hospital) during a period of 10 months.

This double-blinded RCT will include adult patients diagnosed with RA according to the Association of Rheumatology America (ACR) criteria, attending the Rheumatology Department of Charles Nicolle Hospital.

All included patients will be randomized into two groups: an intervention group who will receive omega-3 supplementation and a control group who will receive placebo supplementation, over a period of 3 months.

The placebo capsules will be olive oil-based and will have the same visual as the omega-3 capsules. They will be developed by Vital Company.

Patients in the intervention group will consume 2 omega-3 capsules daily, which contain 36% and 24% of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), respectively.

The dose of omega-3 and placebo will be constant throughout the study period.

Patients will be evaluated at baseline and after 3 months of omega-3 or placebo intake, by a questionnaire performed by a research assistant, which contains the following evaluation parameters:

* Assessment of dietary and non-study supplemental intakes of marine omega-3 fatty acids
* Assessment of disease activity
* Assessment of function
* Assessment of sleep quality
* Assessment of fatigue

DETAILED DESCRIPTION:
Objective:

The aim of this double-blinded randomized controlled trial (RCT) will be to assess the effect of omega-3 intake versus placebo among patients with RA on the primary outcome of disease activity, and the secondary outcomes of function, fatigue and sleep.

Study design This is a prospective, comparative, randomized study, that will be conducted in a single centre (the Rheumatology Department of Charles Nicolle Hospital) during a period of 10 months (from May 2025 to February 2026).

Patients This double-blinded RCT will include adult patients diagnosed with RA according to the Association of Rheumatology America (ACR) criteria, attending the Rheumatology Department of Charles Nicolle Hospital. Concomitant use of synthetic and/or biologic disease modifying antirheumatic drugs (DMARDs) and symptomatic treatments (low dose of corticosteroids, non-steroid anti-inflammatory drugs (NSAIDs)) is permitted by maintaining a stable dose during the study period.

Non-inclusion criteria will be allergy to fish and seafood, treatment with anticoagulants and coagulation disorders, severe hypertriglyceridemia associated with pancreatitis, severe hepatic impairment, severe renal impairment, and current pregnancy or breastfeeding.

Study intervention All included patients will be randomized into two groups: an intervention group who will receive omega-3 supplementation and a control group who will receive placebo supplementation, over a period of 3 months.

The placebo capsules will be olive oil-based and will have the same visual as the omega-3 capsules. They will be developed by Vital Company.

Patients in the intervention group will consume 2 omega-3 capsules daily, which contain 36% and 24% of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), respectively.

The dose of omega-3 and placebo will be constant throughout the study period. Outcome Measures

Patients will be evaluated at baseline and after 3 months of omega-3 or placebo intake, by a questionnaire performed by a research assistant, which contains the following evaluation parameters:

* Assessment of dietary and non-study supplemental intakes of marine omega-3 fatty acids
* Assessment of disease activity
* Assessment of function
* Assessment of sleep quality
* Assessment of fatigue

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years
* Patients diagnosed with RA according to the Association of Rheumatology America (ACR) criteria, attending the Rheumatology Department of Charles Nicolle Hospital.

Exclusion Criteria:

* Patients with allergy to fish and seafood
* Patients treated with anticoagulants and coagulation disorders
* Patients with severe hypertriglyceridemia associated with pancreatitis
* Patients with severe hepatic impairment
* Patients with severe renal impairment
* Current pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
impact of omega3 supplementation on rheumatoid arthritis activity | Rheumatoid arthritis activity will be evaluated at baseline and at the end of the protocol (3 months of supplementation)
  Patients will be evaluated by the disease Activity Score (DAS28). This combined index measures disease activity in patients with RA. It includes a 28 tender joint count, a 28 swollen joint count, a general assessment of the patient's general health status and the level of CRP. The score is interpreted as follow: less than 2.6: RA is in remission, 2.6 to 3.2: a low level of disease activity, more than 3.2: moderate disease activity, more than 5.1: very active disease.

SECONDARY OUTCOMES:
effect of omega3 supplementation on rheumatoid arthritis function | Function in rheumatoid arthrtis will be evaluated at baseline and then 3 months later
  Function will be evaluated by the Health Assessment Questionnaire (HAQ), which is one of the most widely used measures of patient's function, with an acceptable validity and reliability. It contains 8 domains including: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common activities. Each domain is noted 0 to 3 (0=No assistance is needed, 1=A special device is used by the patient in his/her usual activities. 2=The patient usually needs help from another person, 3=The patient usually needs both a special device and help from another person).
  The final score is the sum of the ratings of the various domains divided by the number of domains evaluated. The score obtained in this way is between 0 and 3, with a higher score indicating a higher disability.
effect of omega3 supplementation on fatigue during rheumatoid arthritis | Fatigue will be assessed at baseline, and then 3 months after the omega3 supplementation
  Fatigue will be assessed by the Functional Assessment of Chronic Illness Therapy Fatigue Subscale (FACIT-Fatigue). It is a 13-item measure that assesses physical and functional impact of fatigue. Scores range from 0 to 52, with higher scores indicating less fatigue.
Effect of omega3 supplementation on sleep quality during rheumatoid arthrtis | Sleep quality during rheumatoid arthritis will be assessed at baseline and then 3 months after omega3 supplementation
  Sleep quality will be assessed by the Pittsburgh Sleep Quality Index (PSQI), which is a self-report questionnaire that assesses sleep quality over a one-month time interval. It is composed of 19 items that measure seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping medications and daytime dysfunction. Scores range from 0 to 21, with higher scores indicating poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Charles Nicolle Hospital, Tunis, Bab Saadoun, Tunisia

IPD SHARING:
Plan to Share IPD: No